CLINICAL TRIAL: NCT04245917
Title: Natural History Study of Mitochondrial Neurogastrointestinal Encephalomyopathy
Brief Title: Natural History Study of MNGIE
Status: Suspended | Type: Observational
Why Stopped: Business Reason
Sponsor: Entrada Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ET-NHS-901
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Mitochondrial Neurogastrointestinal Encephalomyopathy
Keywords: MNGIE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MNGIE Patients: Patients with mitochondrial neurogastrointestinal encephalomyopathy
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional natural history study

SUMMARY:
Non-interventional, prospective, multicenter, natural history study of patients with mitochondrial neurogastrointestinal encephalomyopathy (MNGIE)

ELIGIBILITY:
Inclusion Criteria:

* Has MNGIE

Exclusion Criteria:

* Substance abuser

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female MNGIE patients greater than 5 years of age
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
MNGIE Clinical Course | 5 years
  To evaluate the clinical course of MNGIE patients

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Study Chair — Columbia University
Locations (5):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - Columbia University, New York, New York
  - Baylor St Luke's Medical Center and Texas Children's Hospital at Baylor College of Medicine, Houston, Texas
- Turkey (Türkiye) (2):
  - Ege University Medical Faculty; Department of Pediatrics, Bornova, İzmir
  - Gazi Üniversitesi Tıp Fakültesi, Ankara

IPD SHARING:
Plan to Share IPD: No